CLINICAL TRIAL: NCT04799041
Title: Gonyautoxin 2/3 in the Treatment of Acute Back Pain (Study No CLN 17-032): A Clinical Proof-of-concept Study
Brief Title: Gonyautoxin 2/3 in the Treatment of Acute Back Pain: A Clinical Proof-of-concept Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Algenis SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLN 17-032 (Chilean Number)
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Back Pain; Acute Pain
Keywords: Low Back Pain; Acute Pain; Gonyautoxin; Paralytic Shellfish Poison; Muscle Relaxants
MeSH Terms: conditions — Back Pain; Acute Pain; Low Back Pain; Muscle Hypotonia

STUDY DESIGN:
Intervention Model Description: This was a double-blind, placebo-controlled, randomized study in patients with acute back pain. This was a proof of concept study to determine efficacy and safety in two groups: active and placebo. Each patient participated in only one group. This was a single-center clinical trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GTX 2/3 (Active Comparator): Dose level administered of GTX 2/3 was 80 mcg. Dose was administered as IM paravertebral injections, 1 mL per site. Total of 2 mL of GTX 2/3 was injected. The IMP was supplied in glass vials containing 1.2 mL solution at a total GTX 2 and GTX 3 concentration of 40 mcg/mL (at a relative epimer ratio of 62% GTX 2:38% GTX 3).
  Interventions: Drug: GTX 2/3
- Placebo (Placebo Comparator): Placebo was of identical appearance to the IMP, and was administered as IM paravertebral injections, 1 mL per site. Total of 2 mL of placebo was injected.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GTX 2/3 — There were 15 patients in this group. Each one received only one treatment.
  Other Names: NAVX-010 (drug internal name); Gonyautoxin 2/3
  Arms: GTX 2/3
Drug: Placebo — There were 15 patients in this group. Each one received only one treatment.
  Other Names: Placebo of NAVX-010
  Arms: Placebo

SUMMARY:
This was an interventional, double-blind, placebo controlled, randomized, single dose, proof-of-concept study. It was a single-center clinical trial.

The purpose of the study was to explore the clinical efficacy and safety of a single local IM injection of gonyautoxin 2/3 (GTX 2/3) compared to placebo in decreasing pain and improving lumbar functionality at short term follow-up in adult patients with acute low back pain, without radiculopathy.

DETAILED DESCRIPTION:
This was an interventional, double-blind, placebo controlled, randomized, single dose, proof-of-concept study. It was a single-center clinical trial.

The primary objective was to determine the clinical efficacy of GTX 2/3 in the decrease of pain and in the functional improvement of adults patients with acute back pain with no associated radiculopathy. The secondary objective was to determine the safety of a local intramuscular injection of GTX 2/3 in adults patients with acute back pain.

Thirty subjects were studied in 2 groups, each consisting of 15 subjects. One group received the Investigational Medicinal Product (IMP) and the other group received placebo.

The eligible patients were adults, from both sex, aged between 18 and 70 years, with an episode of acute back pain without radiculopathy, with a pain intensity higher than 4 in the VAS scale, with no chronic pain and without any severe pathology.

Each subject participated in 1 treatment group only. All subjects received IV administration of 100 mg Ketoprofen before the IMP injection. All patients returned for a follow-up visit at day 4 after dose administration and at day 7 for discharge. Follow up telephone calls were done on day 1, 2 and 3 after the administration.

Each subject received only a single dose of GTX 2/3 or placebo during the study. Doses were administered as IM paravertebral injections, 1 mL per site. Total of 2 mL of GTX 2/3 or placebo. The IMP was supplied in glass vials containing 1.2 mL solution at a total GTX 2 and GTX 3 concentration of 40 mcg/mL (at a relative epimer ratio of 62% GTX 2:38% GTX 3). The total concentration of drug administrated was 80 mcg. Placebo was of identical appearance to the IMP.

Patients that participated in the study had the possibility of using rescue medication. As a first line medication was Ketoprofen (maximum of 200 mg per day) and as a second line analgesia was Tramadol®.

The primary efficacy endpoints were the mean change in pain intensity and lumbar function from baseline to day 4, as measured by VAS and RMDQ scores, respectively. Secondary outcomes were: 1) the mean change in pain intensity and lumbar function from baseline to day 7 as measured by VAS and RMDQ scores, respectively, 2) the frequency of use of rescue pain drugs during Days 1 to 3, and 3) the occurrence of adverse events during the 7 days of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman patients between 18 and 75 years old.
* Acute back pain episode without radiculopathy asociated and no red flags.
* Back pain related pain bigger than 4 in VAS.
* Patients with no severe illnesses or conditions that would be inappropriate to enroll in this study or patients with no chronic pain.
* Signed informed consent.

Exclusion Criteria:

* Pregnant women or breastfeeding.
* Hyper acute back pain that requires emergency hospitalization.
* Chronic back pain or complicated (red flags).
* Patients that have received previous analgesic therapy of long half life, like corticoids, for current back pain or other pathology (inhalers are excluded).
* Associated neuromuscular diseases, inflammatory diseases in the spine (Musculoskeletal Disorders 2017, 18; 454: 2-12), inability to stand up, tumoral diseases, terminal disease.
* Ongoing local treatment with calcium antagonists or trinitroglycerin.
* Treatment with anti-vitamins K or another anticoagulant.
* Patients with adverse psychosomatic, work or social factors.
* Known or suspected allergy to any component of the study drug.
* Current participation in another clinical study or 30 days prior to enrollment.
* Another condition that in the opinion of the PI prevents participation in the study (physical or mental) or that cannot attend controls or answer the patient's survey / diary.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Efficacy of GTX 2/3 in the treatment of acute back pain after 4 days of administration. | 4 days after one local administration
  Change of pain (0- to 10-point on a Visual Analog Scale (VAS), 0 meaning no pain and 10 the worst pain) and/or functional improvement (0- to 24-point on the Roland-Morris Disability Questionnaire (RMDQ). Each question is one point so scores can range from 0 (no disability) to 24 (severe disability)) in patients with acute back pain without radiculopathy from baseline to day 4 day after one local administration of GTX 2/3 or placebo.

SECONDARY OUTCOMES:
Efficacy of GTX 2/3 in the treatment of acute back pain after 7 days of administration. | 7 days after one local administration
  Change of pain (0- to 10-point on a Visual Analog Scale (VAS), 0 meaning no pain and 10 the worst pain) and/or functional improvement (0- to 24-point on the Roland-Morris Disability Questionnaire (RMDQ). Each question is one point so scores can range from 0 (no disability) to 24 (severe disability)) in patients with acute back pain without radiculopathy from baseline to day 7 day after one local administration of GTX 2/3 or placebo.
Pain evaluation after 2 hours of GTX 2/3 administration (Discharge of the hospital) | 2 hours after one local administration
  Pain evaluation using a Visual Analog Scale (0 no pain and 10 the worst pain) after 2 hours of GTX 2/3 or placebo administration, before the discharge of the patient from the hospital.
Pain evaluation on day 1 after GTX 2/3 administration. | 1 day after one local administration
  Pain evaluation using a Visual Analog Scale (0 no pain and 10 the worst pain) after day 1 of GTX 2/3 or placebo administration.
Pain evaluation on day 2 after GTX 2/3 administration. | 2 day after one local administration
  Pain evaluation using a Visual Analog Scale (0 no pain and 10 the worst pain) after day 2 of GTX 2/3 or placebo administration.
Pain evaluation on day 3 after GTX 2/3 administration. | 3 day after one local administration
  Pain evaluation using a Visual Analog Scale (0 no pain and 10 the worst pain) after day 3 of GTX 2/3 or placebo administration.
Use of rescue medication | 3 days
  Use of rescue medication on day 1, 2 and 3 after GTX 2/3 or placebo administration.
Safety of GTX 2/3 by questioning the patients. | Through the 7 days of the study
  Search of side effects through questioning the patients during all the observation period (7 days). The adverse events questioned included: pain at site injection, perioral paresthesia, limbs paresthesia, headache, nausea, itching at site injection, allergy and ataxia. Indication to notify any event after this period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Bravo, MD, Principal Investigator — Hospital San José
Locations (1):
- Hospital San José SSMN, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No